CLINICAL TRIAL: NCT02920346
Title: Heart Sounds at Home: Prospective Maternal Surveillance of SSA Positive Pregnancies Using a Hand-Held Fetal Heart Rate Monitor
Brief Title: Prospective Maternal Surveillance of SSA (Sjögren Syndrome A) Positive Pregnancies Using a Hand-held Fetal Heart Rate Monitor
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's National Research Institute (Other); Stollery Children's Hospital (Other); The Hospital for Sick Children (Other); New York Presbyterian Hospital (Other); University of California, San Francisco (Other); Children's Hospital of Philadelphia (Other); Karolinska Institutet (Other); St. Justine's Hospital (Other); Johns Hopkins All Children's Hospital (Other); Sanford Health (Other); Seattle Children's Hospital (Other); Eastern Virginia Medical School (Other); Children's Hospital Colorado (Other); University of Minnesota (Other); The University of Texas Health Science Center, Houston (Other); Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 13-1879
Record Dates: First submitted 2016-08-03; First posted 2016-09-30 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Sjogren's Syndrome; Neonatal Systemic Lupus Erythematosus; Fetal Heart Block Complete
Keywords: Neonatal Systemic lupus erythematosus; Sjogren's syndrome; Fetal Atrioventricular Block; Fetal Heart Block
MeSH Terms: conditions — Sjogren's Syndrome; Neonatal Systemic lupus erythematosus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the research study "Heart Sounds at Home" is for pregnant SSA or SSA/SSB (Sjögren syndrome B) antibody positive mothers to use a Doppler fetal heart rate monitor to detect abnormal heart rates and rhythms in their babies before they are born.

DETAILED DESCRIPTION:
The study will enroll mothers during week 16-19 of gestation and will ask the mothers to use a hand-held Doppler monitor to listen to the baby's heart rate and rhythm twice daily from about week 16 to week 26 of the pregnancy. Pregnant mothers will be asked to keep a log of the heart rates and will undergo a fetal echocardiogram every 2 weeks during their study participation. In addition to these procedures, the study team will collect the mother's medical and obstetrical histories. Should irregular heart rhythms be detected at home, the mother will contact the investigator to be evaluated. After the baby is delivered, the study team will collect information about the baby's birth and heart rhythm evaluation (electrocardiogram).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with positive SSA or SSA and SSB antibodies
* Gestational age (GA) between 16 and 19 weeks
* No signs of antibody-mediated fetal cardiac disease on pre-enrollment echo

Exclusion Criteria:

* Subjects who are more than 19 weeks gestation
* Subjects who have a fetus with an estimated fetal weight below the 10th percentile will also not be included

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will include all pregnant women with positive SSA or SSA and SSB antibodies between the gestational ages of 16-19 weeks with no signs of antibody-mediated fetal cardiac disease on pre-enrollment fetal echocardiogram. Subjects who are more than 19 weeks gestation will not be included. Subjects who have a fetus with an estimated fetal weight below the 10th percentile will also not be included.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Development of Fetal AV (atrio-ventricular) heart block | Date of randomization until the date of first documented progression, assessed up to 41 weeks.
  Development of fetal AV heart block will be determined by the principal investigator's analysis of the fetal echocardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina F Cuneo, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuneo BF, Strasburger JF, Niksch A, Ovadia M, Wakai RT. An expanded phenotype of maternal SSA/SSB antibody-associated fetal cardiac disease. J Matern Fetal Neonatal Med. 2009 Mar;22(3):233-8. doi: 10.1080/14767050802488220. PMID 19330707
- [Background] Cuneo BF, Lee M, Roberson D, Niksch A, Ovadia M, Parilla BV, Benson DW. A management strategy for fetal immune-mediated atrioventricular block. J Matern Fetal Neonatal Med. 2010 Dec;23(12):1400-5. doi: 10.3109/14767051003728237. Epub 2010 Apr 12. PMID 20384469
- [Derived] Cuneo BF, Sonesson SE, Levasseur S, Moon-Grady AJ, Krishnan A, Donofrio MT, Raboisson MJ, Hornberger LK, Van Eerden P, Sinkovskaya E, Abuhamad A, Arya B, Szwast A, Gardiner H, Jacobs K, Freire G, Howley L, Lam A, Kaizer AM, Benson DW, Jaeggi E. Home Monitoring for Fetal Heart Rhythm During Anti-Ro Pregnancies. J Am Coll Cardiol. 2018 Oct 16;72(16):1940-1951. doi: 10.1016/j.jacc.2018.07.076. PMID 30309472
- See also: study website — http://www.heartsoundsathome.com